CLINICAL TRIAL: NCT00674583
Title: Non-inferiority of GSK Biologicals' Meningococcal Vaccine (GSK134612) Compared to Licensed MenC-CRM197 Conjugate Vaccine in Healthy Children
Brief Title: Comparison of GSK Biologicals' Meningococcal Vaccine (GSK134612) and Licensed MenC-CRM197 Vaccine in Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111414; 2007-007837-38 (EudraCT Number)
Record Dates: First submitted 2008-05-07; First posted 2008-05-08 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Infections, Meningococcal
Keywords: Conjugate vaccine; Meningococcal disease; Immunogenicity; Meningococcal vaccine; Safety
MeSH Terms: conditions — Meningococcal Infections

ARMS (2):
- Nimenrix Group (Experimental): Healthy male or female subjects between, and including 2 and 10 years of age, intramuscularly received 1 dose of Nimenrix™ vaccine into the non-dominant deltoid region, at Day 0.
  Interventions: Biological: GSK Biologicals' meningococcal vaccine GSK134612
- Menjugate Group (Active Comparator): Healthy male or female subjects between, and including 2 and 10 years of age, intramuscularly received 1 dose of Menjugate® vaccine into the non-dominant thigh region, at Day 0.
  Interventions: Biological: Menjugate

INTERVENTIONS:
Biological: GSK Biologicals' meningococcal vaccine GSK134612 — Intramuscular administration, 1 dose
  Arms: Nimenrix Group
Biological: Menjugate — Intramuscular administration, 1 dose
  Other Names: MenC-CRM197vaccine
  Arms: Menjugate Group

SUMMARY:
The purpose of the study is to investigate whether or not GSK Biologicals' meningococcal vaccine GSK134612 is inferior to a licensed MenC-CRM197 conjugate vaccine in terms of vaccine antibody response against meningococcal serogroup C disease.

DETAILED DESCRIPTION:
The study has 2 study groups. One group will receive one dose of GSK Biologicals' vaccine GSK 134612 and the other group will receive one dose of licensed MenC-CRM197 vaccine. All subjects will have 2 blood samples taken: just before vaccination and one month after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose parents/guardians, the investigator believes can and will comply with the requirements of the protocol.
* A male or female between, and including, 2 and 10 years of age at the time of the vaccination.
* Written informed consent obtained from the parent(s) or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Previously completed routine childhood vaccinations to the best of his/her parents'/guardians' knowledge.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the study vaccine dose, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose..
* Administration of a vaccine not foreseen by the study protocol during the period starting from one month before the dose of the study vaccine and ending 30 days after.
* Concurrently participating in another clinical study or planned participation in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous vaccination with meningococcal polysaccharide vaccine of serogroup A, C W-135 and/or Y (for subjects below 6 years) or within the last five years (for subjects 6 years old and above).
* Previous vaccination with meningococcal polysaccharide conjugate vaccine serogroups A, C, W-135 and/or Y.
* History of meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment
* Administration of immunoglobulins and/or any blood products within the three months preceding the study vaccine dose or planned administration during the study period.

Exclusion criteria for specified regions in France

* Subjects in contact with somebody suffering from an invasive infection with meningococcal serogroups A, C, Y or W-135, or
* Subjects living in a geographic area in France where local outbreak with meningococcal serogroup C has occurred and would thus be likely to participate in a vaccination campaign against meningococcal serogroup C.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 414 (Actual)
Dates: Start 2008-05-09 (Actual); Primary Completion 2008-09-02 (Actual); Study Completion 2009-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (27):
- France (11):
  - GSK Investigational Site, Draguignan
  - GSK Investigational Site, Laon
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Lingolsheim
  - GSK Investigational Site, Miribel
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Laurent-du-Var
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Vaulx-en-Velin
  - GSK Investigational Site, Vence
- Germany (16):
  - GSK Investigational Site, Tettnang, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Espelkamp, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Heiligenhaus, North Rhine-Westphalia
  - GSK Investigational Site, Hille, North Rhine-Westphalia
  - GSK Investigational Site, Porta Westfalica, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Velbert, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Knuf M, Romain O, Kindler K, Walther U, Tran PM, Pankow-Culot H, Fischbach T, Kieninger-Baum D, Bianco V, Baine Y, Miller J. Immunogenicity and safety of the quadrivalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine (MenACWY-TT) in 2-10-year-old children: results of an open, randomised, controlled study. Eur J Pediatr. 2013 May;172(5):601-12. doi: 10.1007/s00431-012-1924-0. Epub 2013 Jan 11. PMID 23307281
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 111414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria,contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | Nimenrix Group | Menjugate Group
Started | 311 | 103
Completed | 311 | 103
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix Group | Menjugate Group | Total
Number analyzed (Participants) | 311 | 103 | 414
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.6 (2.52) | 5.6 (2.32) | 5.6 (2.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 51 | 214
  Male | 148 | 52 | 200
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 13 | 6 | 19
  Asian-Central/South Asian heritage | 1 | 0 | 1
  Asian-East Asian heritage | 2 | 1 | 3
  Asian-Japanese heritage | 1 | 0 | 1
  Asian-South East Asian heritage | 3 | 1 | 4
  White-Arabic/North African heritage | 16 | 6 | 22
  White-Caucasian/European heritage | 267 | 87 | 354
  Not specified | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Vaccine Response to Meningococcal Serogroup C Serum Based on a Bactericidal Assay Using Baby Rabbit Complement (rSBA-MenC) Antibody
Description: Vaccine response to MenC was defined as: -for initially seronegative subjects [i.e. rSBA-MenC titer below (<) 1:8], antibody titer greater than or equal to (≥) 1:32; -for initially seropositive (i.e. rSBA-MenC titer ≥ 1:8), antibody titer post-vaccination ≥ 4-fold the pre-vaccination antibody titer.
Time Frame: One month after vaccination (Month 1)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures and assay results for antibodies against at least one study vaccine antigen component after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 268 | 92
Participants | 254 | 88
Statistical Analysis 1: Comparison: Nimenrix Group vs Menjugate Group; To demonstrate the non-inferiority of the Nimenrix group compared to the Menjugate group, two-sided standardized asymptotic 95% confidence interval (CI) for the groups difference [Nimenrix group minus Menjugate group] in the percentages of subjects with bactericidal vaccine response to MenC was computed; Test type: Non-Inferiority — Criterion for non-inferiority evaluation: The lower limit (LL) of the two-sided standardized asymptotic 95% CI for the group difference (Nimenrix Group minus Menjugate Group) in the percentages of subjects with vaccine response to rSBA-MenC is greater than or equal to (≥) the pre-defined clinical limit of -10%; Difference in percentage = -0.88, 95% CI 2-sided [-5.25 to 5.75]

2. Secondary Outcome: Meningococcal Serogroup A (rSBA) Antibody Titers by Serogroup
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Prior to (Month 0) and one month after vaccination (Month 1)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures and assay results for antibodies against at least one study vaccine antigen component after vaccination were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 296 | 97
Titers
  rSBA-MenA, Month 0: number analyzed (Participants) | 227 | 76
  rSBA-MenA, Month 0 | 31.5 [23.3 to 42.5] | 25.9 [15.6 to 43]
  rSBA-MenA, Month 1: number analyzed (Participants) | 294 | 82
  rSBA-MenA, Month 1 | 6236.1 [5574.5 to 6976.3] | 27.2 [15.6 to 47.4]
  rSBA-MenC, Month 0: number analyzed (Participants) | 270 | 94
  rSBA-MenC, Month 0 | 22.7 [18.1 to 28.4] | 19.4 [13.1 to 28.8]
  rSBA-MenC, Month 1: number analyzed (Participants) | 293 | 97
  rSBA-MenC, Month 1 | 2794.8 [2393.5 to 3263.3] | 5291.6 [3814.6 to 7340.5]
  rSBA-MenW-135, Month 0: number analyzed (Participants) | 282 | 92
  rSBA-MenW-135, Month 0 | 83.2 [67.9 to 102] | 70.2 [48.5 to 101.6]
  rSBA-MenW-135, Month 1: number analyzed (Participants) | 296 | 95
  rSBA-MenW-135, Month 1 | 8549.5 [7618.5 to 9594.3] | 87.3 [58.5 to 130.4]
  rSBA-MenY, Month 0: number analyzed (Participants) | 285 | 90
  rSBA-MenY, Month 0 | 153.6 [125.3 to 188.3] | 107.4 [71.4 to 161.6]
  rSBA-MenY, Month 1: number analyzed (Participants) | 295 | 95
  rSBA-MenY, Month 1 | 8360.7 [7447.3 to 9386.1] | 128.2 [83.8 to 196.2]

3. Secondary Outcome: Anti-meningococcal Serogroup Polysaccharides (Anti-PS) Antibody Concentrations
Description: Anti-PSA, anti-PSC, anti-PSW-135 and anti-PSY antibody concentrations were presented as geometric mean concentrations (GMCs) and tabulated as micrograms per milliliter (μg/mL).
Time Frame: Prior to (Month 0) and one month after vaccination (Month 1)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 149 | 52
μg/mL
  Anti-PSA, Month 0: number analyzed (Participants) | 148 | 52
  Anti-PSA, Month 0 | 0.2 [0.17 to 0.22] | 0.22 [0.17 to 0.29]
  Anti-PSA, Month 1: number analyzed (Participants) | 149 | 50
  Anti-PSA, Month 1 | 32.45 [26.57 to 39.63] | 0.31 [0.19 to 0.49]
  Anti-PSc, Month 0: number analyzed (Participants) | 147 | 52
  Anti-PSc, Month 0 | 0.18 [0.16 to 0.2] | 0.2 [0.16 to 0.25]
  Anti-PSc, Month 1 | 14.95 [12.89 to 17.34] | 18.07 [13.88 to 23.51]
  Anti-PSW-135, Month 0: number analyzed (Participants) | 144 | 47
  Anti-PSW-135, Month 0 | 0.17 [0.15 to 0.18] | 0.17 [0.14 to 0.2]
  Anti-PSW-135, Month 1: number analyzed (Participants) | 144 | 47
  Anti-PSW-135, Month 1 | 6.96 [5.72 to 8.47] | 0.18 [0.15 to 0.22]
  Anti-PSY, Month 0: number analyzed (Participants) | 147 | 47
  Anti-PSY, Month 0 | 0.16 [0.15 to 0.17] | 0.16 [0.15 to 0.17]
  Anti-PSY, Month 1: number analyzed (Participants) | 144 | 47
  Anti-PSY, Month 1 | 14.15 [11.66 to 17.17] | 0.17 [0.15 to 0.19]

4. Secondary Outcome: Number of Subjects Between 2 and 5 Years of Age With Any and Grade 3 Solicited Local Symptoms
Description: Solicited symptoms assessed were: pain, redness and swelling. Any = occurrence of any local symptom regardless of their intensity grade. Grade 3 Pain = cried when limb was moved/spontaneously painful. Grade 3 Redness and Swelling= redness/swelling spreading beyond (>) 30 millimeters (mm).
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with their symptom sheets filled in, for whom data were available.
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix Group (< 6 Years): Healthy male or female subjects between, and including 2 to 5 years of age, intramuscularly received 1 dose of Nimenrix™ vaccine into the non-dominant deltoid region, at Day 0.
- Menjugate Group (< 6 Years): Healthy male or female subjects between, and including 2 to 5 years of age, intramuscularly received 1 dose of Menjugate® vaccine into the non-dominant thigh region, at Day 0.
Arm/Group | Nimenrix Group (< 6 Years) | Menjugate Group (< 6 Years)
Number analyzed (Participants) | 162 | 53
Participants
  Any Pain | 45 | 15
  Grade 3 Pain | 0 | 1
  Any Redness | 57 | 21
  Grade 3 Redness | 11 | 8
  Any Swelling | 43 | 13
  Grade 3 Swelling | 7 | 3

5. Secondary Outcome: Number of Subjects Between 6 and 10 Years of Age With Any and Grade 3 Solicited Local Symptoms
Description: Solicited symptoms assessed were: pain, redness and swelling. Any = occurrence of any local symptom regardless of their intensity grade. Grade 3 Pain = pain that prevented normal activity. Grade 3 Redness and Swelling= redness/swelling spreading beyond (>) 50 millimeters (mm).
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix Group (≥ 6 Years): Healthy male or female subjects between, and including 6 and 10 years of age, intramuscularly received 1 dose of Nimenrix™ vaccine into the non-dominant deltoid region, at Day 0.
- Menjugate Group (≥ 6 Years): Healthy male or female subjects between, and including 6 and 10 years of age, intramuscularly received 1 dose of Menjugate® vaccine into the non-dominant thigh region, at Day 0.
Arm/Group | Nimenrix Group (≥ 6 Years) | Menjugate Group (≥ 6 Years)
Number analyzed (Participants) | 148 | 50
Participants
  Any Pain | 65 | 27
  Grade 3 Pain | 3 | 3
  Any Redness | 58 | 19
  Grade 3 Redness | 9 | 5
  Any Swelling | 44 | 15
  Grade 3 Swelling | 4 | 3

6. Secondary Outcome: Number of Subjects Between 2 and 5 Years of Age With Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed were drowsiness, fever [defined as oral temperature ≥ 37.5 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of the general symptom regardless of intensity grade and relationship to vaccination. Grade 3 Symptom = symptom that prevented normal activity. Grade 3 Loss of appetite = did not eat at all. Grade 3 Fever = fever > 39.5°C. Related = general symptoms assessed by the investigator as causally related to vaccination
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group (< 6 Years) | Menjugate Group (< 6 Years)
Number analyzed (Participants) | 162 | 53
Participants
  Any Drowsiness | 23 | 6
  Grade 3 Drowsiness | 0 | 1
  Related Drowsiness | 15 | 6
  Any Fever | 9 | 3
  Grade 3 Fever | 0 | 0
  Related Fever | 9 | 3
  Any Irritability | 25 | 6
  Grade 3 Irritability | 1 | 1
  Related Irritability | 16 | 5
  Any Loss of appetite | 17 | 5
  Grade 3 Loss of appetite | 0 | 0
  Related Loss of appetite | 9 | 4

7. Secondary Outcome: Number of Subjects Between 6 and 10 Years of Age With Any, Grade 3 and Related Solicited General Symptoms
Description: as for outcome 6
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group (≥ 6 Years) | Menjugate Group (≥ 6 Years)
Number analyzed (Participants) | 148 | 50
Participants
  Any Fatigue | 33 | 11
  Grade 3 Fatigue | 4 | 0
  Related Fatigue | 29 | 7
  Any Fever (Orally) | 10 | 1
  Grade 3 Fever (Orally) | 0 | 0
  Related Fever (Orally) | 9 | 0
  Any Gastrointestinal | 22 | 4
  Grade 3 Gastrointestinal | 1 | 0
  Related Gastrointestinal | 13 | 3
  Any Headache | 30 | 4
  Grade 3 Headache | 2 | 0
  Related Headache | 24 | 2

8. Secondary Outcome: Number of Subjects Reporting Specific Adverse Events
Description: Specific AEs included: - rash (hives, idiopathic thrombocytopenic purpura, petechiae); - new onset of chronic illness(es) (NOCI) (e.g. autoimmune disorders, asthma, type I diabetes and allergies); - conditions prompting emergency room (ER) visits.
Time Frame: Up to 6 months after vaccination (Month 6)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 311 | 103
Participants
  Any Rash(es) | 8 | 1
  Any NOCI(s) | 1 | 1
  Any ER visit(s) | 11 | 1

9. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 311 | 103
Participants | 55 | 20

10. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Up to six months after vaccination (Month 6)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 311 | 103
Participants | 6 | 1

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 4-day (Days 0-3) post-vaccination period. Unsolicited adverse events (AEs): during the 31-day (Days 0-30) post-vaccination period. Serious adverse events (SAEs): from Day 0 up to Month 6 post-vaccination.
Description: The solicited local and general symptoms were only collected from those subjects who filled in their symptom sheets.
Arm/Group | Nimenrix Group | Menjugate Group
All-Cause Mortality (participants affected / at risk) | 0/311 | 0/103
Serious Adverse Events (participants affected / at risk) | 6/311 | 1/103
Other Adverse Events (participants affected / at risk) | 181/311 | 63/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix Group (N=311) | Menjugate Group (N=103)
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0
Accidental poisoning (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nimenrix Group (N=311) | Menjugate Group (N=103)
Pain (General disorders) | 110/310 | 42
Redness (General disorders) | 115/310 | 40
Swelling (General disorders) | 87/310 | 28
Drowsiness (< 6 years) (General disorders) | 23/162 | 6/53 — This solicited general symptom was assessed for subjects between 2 to 5 years of age, from the two groups.
Fever (General disorders) | 19/310 | 4
Irritability (< 6 years) (General disorders) | 25/162 | 6/53 — This solicited general symptom was assessed only for subjects between 2 to 5 years of age, from the two groups.
Loss of appetite (< 6 years) (General disorders) | 17/162 | 5/53 — This solicited general symptom was assessed only for subjects between 2 to 5 years of age, from the two groups.
Fatigue (≥ 6 years) (General disorders) | 33/148 | 11/50 — This solicited general symptom was assessed only for subjects between 6 to 10 years of age, from the two groups.
Gastrointestinal (≥ 6 years) (General disorders) | 22/148 | 4/50 — This solicited general symptom was assessed only for subjects between 6 to 10 years of age, from the two groups.
Headache (≥ 6 years) (General disorders) | 30/148 | 4/50 — This solicited general symptom was assessed only for subjects between 6 to 10 years of age, from the two groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.